CLINICAL TRIAL: NCT03088410
Title: The Tshilo Dikotla Study: Metabolic Outcomes of Children HIV/ARV-Exposed Uninfected in Botswana (MOCHA)
Brief Title: Study of HIV-Infected and Uninfected Pregnant Woman/Child Dyads in Gaborone, Botswana
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jennifer Jao, Associate Professor, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB 2019-2922; R01DK109881 (NIH); HRDC 00781 (Other: Botswana MOH - Health Research Development Committee)
Record Dates: First submitted 2017-03-03; First posted 2017-03-23 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: HIV; Insulin Sensitivity; Diabetes Mellitus
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus | interventions — Zidovudine; Nevirapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Single blind - one party, either the investigator or participant, is unaware of the intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Nevirapine (Experimental): 150 HIV-Exposed Uninfected (HEU) infants on Nevirapine (NVP) Prophylaxis
  Interventions: Drug: Nevirapine
- Zidovudine (Active Comparator): 150 HIV-Exposed Uninfected (HEU) infants on Zidovudine (AZT) Prophylaxis
  Interventions: Drug: Zidovudine
- HIV- unexposed Uninfected (HUU) Infants (No Intervention): 150 HIV- unexposed Uninfected (HUU) Infants

INTERVENTIONS:
Drug: Zidovudine — neonatal 4 weeks prophylactic
  Other Names: AZT
  Arms: Zidovudine
Drug: Nevirapine — neonatal 4 weeks prophylactic
  Other Names: NVP
  Arms: Nevirapine

SUMMARY:
The purpose of this study is to assess the early longitudinal metabolic effects including insulin sensitivity in HIV-exposed uninfected (HEU) children compared to HIV-unexposed uninfected (HUU) children; as well as to determine differences in the effects of neonatal zidovudine (AZT) vs. nevirapine (NVP) prophylaxis on early longitudinal changes in insulin sensitivity in the first 3 years of life.

DETAILED DESCRIPTION:
This study will consist of a nested randomized component of HIV-infected (HIV+) and -uninfected (HIV-) pregnant woman/child dyads in Botswana which will take place in Gaborone, Botswana at Botswana-Harvard AIDS Institute Partnership's (BHPs) clinical research facilities. A total of 300 HIV+ pregnant woman/fetus dyads on cART and 150 HIV- pregnant woman/fetus dyads will be evaluated for insulin sensitivity and followed through the child's 3rd birthday. Amongst HEU infants, participants will be randomized at birth 1:1 with 150 to receive neonatal AZT prophylaxis and 150 to receive neonatal NVP prophylaxis. Targeted metabolomics will be used to assess the role intermediary metabolites in insulin resistance and directly assess mitochondrial function using Seahorse XF96e technology. At the time of study enrollment, all women must be willing to exclusively breastfeed for the infant's first 6 months of life. If in utero and neonatal HIV/ARV exposures are found to be associated with derangements in intermediary metabolism such that HEU infants are at increased risk for insulin resistance by 3 years of age, this would impact screening and prevention strategies for diabetes in this vulnerable population and argue for further research to identify prenatal and neonatal ARV regimens with superior PMTCT efficacy but minimal adverse metabolic consequences.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected and uninfected pregnant women between 16-36 weeks GA are eligible for study enrollment.
* Women must be 18 years of older and able to provide informed consent for themselves and their infant to participate in the study.
* Participants must be Botswana citizens.
* Women must have evidence of HIV infection status. Women NOT documented as HIV seropositive must have documentation of HIV seronegativity during the present pregnancy at or after 32 weeks GA. Women who have an initial negative HIV test during the present pregnancy which was done at <32 weeks GA will need to undergo repeat testing on or after 32 weeks GA in accordance with national guidelines.
* HIV-uninfected women must be willing to undergo HIV pre-test counseling, rapid HIV testing and post-test counseling, referred to as HIV Testing and Counseling (HTC) during pregnancy.
* Women must be willing to remain in study area with their infant and attend scheduled study visits as described above until the child's 3rd birthday.
* For HIV-infected women, they must be on TDF/3TC or FTC/EFV or TDF/3TC or FTC/Dolutegravir at time of study enrollment or willing to initiate this treatment and continue throughout the period of breastfeeding, if not for their lifetime.
* At enrollment, all women must be willing to breastfeed exclusively for the first six months of life.

Exclusion Criteria:

•Pre-existing maternal diabetes mellitus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Homeo-static Model Assessment-Insulin Resistance (HOMA-IR) | up to 3 years
  [glucose (mg/dL) X insulin ( μU/mL)405]

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Jao, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Botswana-Harvard AIDS Institute Partnership, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banda FM, Powis KM, Sun S, Makhema J, Masasa G, Yee LM, Jao J. Fetal biometry following in-utero exposure to dolutegravir-based or efavirenz-based antiretroviral therapy. AIDS. 2020 Dec 1;34(15):2336-2337. doi: 10.1097/QAD.0000000000002674. No abstract available. PMID 32910067
- [Derived] Jao J, Sun S, Bonner LB, Legbedze J, Mmasa KN, Makhema J, Mmalane M, Kgole S, Masasa G, Moyo S, Gerschenson M, Mohammed T, Abrams EJ, Kurland IJ, Geffner ME, Powis KM. Lower Insulin Sensitivity in Newborns With In Utero HIV and Antiretroviral Exposure Who Are Uninfected in Botswana. J Infect Dis. 2022 Nov 28;226(11):2002-2009. doi: 10.1093/infdis/jiac416. PMID 36240387